CLINICAL TRIAL: NCT02994381
Title: A Phase I, Single-Centre, Single Dose Oral Excretion Balance Study of [14C]-RPC1063 in Healthy Male Adults
Brief Title: A Single Dose Oral Excretion Balance Study of [14C]-RPC1063 in Healthy Male Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RPC01-1909
Record Dates: First submitted 2016-12-13; First posted 2016-12-15 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Healthy Volunteers
Keywords: Healthy Male Adults; 14C; RPC1063
MeSH Terms: interventions — ozanimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [14C]-RPC1063 Solution (0.1 g/mL) (Experimental): 1 mg; 10 mL [14C]-RPC1063 HCl oral dose containing NMT 1.3 MBq (37 μCi) 14C
  Interventions: Drug: RPC1063

INTERVENTIONS:
Drug: RPC1063

SUMMARY:
This will be an open-label, non-randomized, single oral dose study in healthy male subjects.

All subjects will receive a single oral dose of 10 mL of [14C]-RPC1063 Solution (0.1 mg/mL), containing NMT 1.3 MBq (37 μCi) 14C.

DETAILED DESCRIPTION:
Subjects will be screened for eligibility to participate in the study up to 28 days before dosing. Subjects will be admitted to the clinical unit on the morning of Day -1 prior to IMP administration. Subjects will be dosed on the morning of Day 1 following a standard breakfast, and will remain resident in the clinic until up to 168 h after dosing. It is planned that subjects will be released as a group when all subjects have achieved a mass balance cumulative recovery of >90% or if <1% of the dose administered has been collected in urine and faeces within 2 separate, consecutive 24 h periods. This may be earlier than 168 h post-dose but no sooner than 96 h post-dose. In this case, collection of all samples (blood, urine and faeces) will be stopped and the subjects will undergo discharge assessments. If this criteria has not been met by all subjects on Day 8, home collections of urine and faeces may be requested at the discretion of the investigator for individual subjects. A follow-up phone call will take place 5 to 10 days after discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male
2. Subject is 30 to 65 years of age
3. Subject has a body weight of at least 50 kg; body mass index (BMI) of 18.0 to 32.0 kg/m2 or, if outside the range, considered not clinically significant by the investigator
4. Subject is willing and able to communicate and participate in the whole study
5. Subject has regular bowel movements (average stool production ≥1 and ≤3 stools per day)
6. Subject has suitable veins for multiple cannulation as assessed by the investigator at screening
7. Subject is able to comprehend the informed consent form, provide written informed consent, and able to comply with requirements of the study.
8. Subject agrees to use an adequate method of contraception

Exclusion Criteria:

1. Subject has received any investigational medicinal product (IMP) in a clinical research study within the previous 3 months
2. Subject is a study site employee or an immediate family member of a study site or sponsor employee
3. Subject has a history of any drug or alcohol abuse in the past 2 years
4. Subject has regular alcohol consumption of >21 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
5. Subject is a current smoker or has smoked within the last 12 months; including cigarettes, e-cigarettes and nicotine replacement products. Positive cotinine test result at screening and admission
6. Subject has radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 millisievert (mSv) in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study
7. Subjects has been enrolled in an absorption, distribution, metabolism and elimination (ADME) study in the last 12 months
8. Subject has clinically significant abnormal biochemistry or haematology as judged by the investigator
9. Subject has positive drugs of abuse test result
10. Subject has positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
11. Subject has evidence of renal impairment at screening and admission, as indicated by an estimated creatinine clearance (CLcr) of <90 mL/min using the Cockcroft-Gault equation
12. Subject has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) concentration >1.25 × the ULN at screening
13. Subject has history of cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease as judged by the investigator
14. Subject has had serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
15. Subject has presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active
16. Subject has donated or lost greater than 400 mL of blood within the previous 3 months
17. Subject is taking, or has taken, any prescribed or over-the-counter drug (other than 2 g per 24 h paracetamol) dietary or herbal remedies within 14 days before IMP administration, or has taken St. John's wort within 28 days before IMP administration. Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the PI and sponsor's medical monitor.
18. Subject fails to satisfy the investigator of fitness to participate for any other reason

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Percentage of elimination of [14C]-RPC1063 | Up to 4 weeks
  Total recovery of radioactivity in urine and feces expressed as a percentage of total radioactive dose in each 24 h interval and cumulatively
Pharmacokinetic- amount of drug excreted | Up to 4 weeks
  Cumulative amount of drug excreted unchanged in the drug in urine

SECONDARY OUTCOMES:
Pharmacokinetic- Cmax | Up to 8 days
  Maximum observed concentration
Pharmacokinetic- Tmax | Up to 8 days
  Time at maximum observed concentration
Pharmacokinetic- AUC0-last | Up to 8 days
  Area under the curve from 0 time to last measurable concentration
Pharmacokinetic- AUC0-inf | Up to 8 days
  Area under the curve from 0 time extrapolated to infinity
Pharmacokinetic- λz | Up to 8 days
  Elimination rate constant
Pharmacokinetic- t1/2 | Up to 8 days
  Terminal elimination half-life
Pharmacokinetic- CL/F | Up to 8 days
  Clearance, the apparent volume cleared of parent drug per unit time after extravascular administration
Pharmacokinetic- Vz/F | Up to 8 days
  The apparent volume of distribution after extravascular administration
Pharmacokinetic- CLr | Up to 8 days
  Renal clearance
Adverse Events (AEs) | Approximately 2 months
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Tran, Pharm.D, Study Director — Celgene Corporation
Locations (1):
- Quotient Clinical, Nottingham, United Kingdom